CLINICAL TRIAL: NCT04931368
Title: Optimizing MATRix as Remission Induction in PCNSL: De-escalated Induction Treatment in Newly Diagnosed Primary CNS Lymphoma - a Randomized Phase III Trial
Brief Title: OptiMATe: De-escalated Induction Treatment in Primary CNS Lymphoma
Acronym: OptiMATe
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Klinikum Stuttgart (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCC215
Record Dates: First submitted 2020-08-25; First posted 2021-06-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Primary Central Nervous System Lymphoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control treatment (Arm A) (Active Comparator): Patients receive four courses of MATRix (Rituximab 2 x 375 mg/m2, HD-Methotrexate 3.5 g/m2, HD-Cytarabine 2 x 2 g/m2, Thiotepa 30 mg/m2; i.v.) as induction treatment. Response assessment with gadolinium-enhanced brain MRI (centrally reviewed) takes place after course two and four. Patient with at least PR proceed to 3rd course of MATRix after first response assessment and to HCT-ASCT (BCNU 400 mg/m2, Thiotepa 4 x 5 mg/kg; i.v.) after second response assessment. Collection of autologous stem cells is planed after the second course of MATRix.
  Interventions: Drug: Control intervention: four courses of MATRix
- Experimental treatment (Arm B) (Experimental): As induction treatment, patients receive one course of Rituximab/HD-Methotrexate (Rituximab 375 mg/m2, HD-Methotrexate 3.5 g/m2; i.v.). In the absence of clinical signs of progression, patients proceed to two courses of MATRix (Rituximab 2 x 375 mg/m2, HD-Methotrexate 3.5 g/m2, HD-Cytarabine 2 x 2 g/m2, Thiotepa 30 mg/m2; i.v.) followed by a response assessment with gadolinium-enhanced brain MRI (centrally reviewed). Patients with at least PR will proceed to HCT-ASCT (BCNU 400 mg/m2, thiotepa 4 x 5 mg/kg; i.v.). Collection of autologous stem cells is planed after the first course of MATRix
  Interventions: Drug: Experimental Treatment: one course Rituximab/HD-Methotrexate, two courses of MATRix

INTERVENTIONS:
Drug: Experimental Treatment: one course Rituximab/HD-Methotrexate, two courses of MATRix — De-escalated induction treatment with R/HD-MTX and two courses of MATRix
  Arms: Experimental treatment (Arm B)
Drug: Control intervention: four courses of MATRix — Patients receive four courses of MATRix as induction treatment.
  Arms: Control treatment (Arm A)

SUMMARY:
This phase III study investigates if a de-escalated induction treatment in newly diagnosed primary CNS lymphoma is superior to the standard MATRix protocol in terms of event free survival.

DETAILED DESCRIPTION:
This phase III study investigates if a de-escalated induction treatment in newly diagnosed primary CNS lymphoma is superior to the standard MATRix protocol in terms of event free survival. Two arms are compared, in the experimental treatment group, participants receive one course of R/HD-MTX, followed by two courses of MATRix and autologous stem cell transplantation. In the control treatment, participants receive four coourses of MATRix followed by autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Immunocompetent patients with newly diagnosed primary diffuse large B-cell lymphoma of the central nervous system (PCNSL).
2. Male or female patients aged 18-65 years irrespective of ECOG or 66-70 years with ECOG Performance Status ≤2.
3. Histologically or cytologically assessed diagnosis of B-cell lymphoma by local pathologist. Diagnostic sample obtained by stereotactic or surgical biopsy, CSF cytology examination or vitrectomy.
4. Disease exclusively located in the CNS.
5. At least one measurable lesion.
6. Previously untreated patients (previous or ongoing steroid treatment admitted)
7. Negative pregnancy test
8. Written informed consent obtained according to international guidelines and local laws by patient or authorized legal representative in case patient is temporarily legally not competent due to his or her disease.
9. Ability to understand the nature of the trial and the trial related procedures and to comply with them.

Exclusion Criteria:

1. Congenital or acquired immunodeficiency including HIV infection and previous organ transplantation.
2. Systemic lymphoma manifestation (outside the CNS).
3. Primary vitreoretinal lymphoma without manifestation in the brain parenchyma or spinal cord
4. Previous or concurrent malignancies with the exception of surgically cured carcinoma in situ of the cervix, carcinoma of the skin or other kinds of cancer without evidence of disease for at least 5 years.
5. Previous Non-Hodgkin lymphoma at any time.
6. Inadequate renal function (clearance < 60 ml/min).
7. Inadequate bone marrow, cardiac, pulmonary or hepatic function according to investigator´s decision
8. Active hepatitis B or C disease.
9. Concurrent treatment with other experimental drugs or participation in an interventional clinical trial with study medication being administered within the last 30 days before the start of this study.
10. Third space fluid accumulation > 500 ml.
11. Hypersensitivity to study treatment or any component of the formulation.
12. Taking any medications that are likely to cause interactions with the study medication
13. Known or persistent abuse of medication, drugs or alcohol.
14. Active COVID-19-infection or non-compliance with the prevailing hygiene measures regarding the COVID-19 pandemic
15. Patients without legal capacity who are unable to understand the nature, significance and consequences of the trial and without designated legal representative.
16. Previous participation in this trial.
17. Persons who are in a relationship of dependency/employment with the sponsor and/or the investigator.
18. Any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
19. Current or planned pregnancy, nursing period
20. For fertile patients: Failure to use one of the following safe methods of contraception: intra-uterine device or hormonal contraception in combination with a mechanical method of contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | up to 24 months after end of treatment
  time from randomization to premature end of treatment due to any reason, lymphoma progression or death, whichever occurs first

SECONDARY OUTCOMES:
Overall survival (OS) | up to 24 months after end of treatment
  time from randomization to death of any course
Progression free survival (PFS) | up to 24 months after end of treatment
  time from randomization until disease progression, relapse or death from any cause
Remission rate prior to consolidation therapy | assesed at RA II (Arm B: day 18-20 of cycle 2, each cycle is 21 days. Arm A: day 18-20 of cycle 4, each cycle is 21 days)
  Remission prior to consolidation therapy will be determined at RA II and will be divided in CR, uCR, PR, CD, PD according to IPCG criteria
Remission rate after consolidation therapy | 30 days after ASCT
  Remission after consolidation therapy will be determined on day 30 after ASCT and will be divided in CR, uCR, PR, SD, PD according to IPCG criteria
rate of patients reaching consolidation therapy | determined up to 4 weeks after response assessment II
  defined as obtaining at least the first dose of consolidation therapy, will be determined after the response assessment II (following 4 cycles of MATRix in the control arm and following 1 cycle of R/HD-MTX and 2 cycles of MATRix in the experimental arm)
Quality of life (QOL), EORTC QLQ-C30, | up to 24 months after end of treatment
  EORTC (European Organization for research and cancer treatment) QLQ-C30, measured during screening, at response assessment II, and with beginning of RA III every 12 months until end of follow-up
Quality of life (QOL), QLQ-BN20 | up to 24 months after end of treatment
  EORTC (European Organization for research and cancer treatment) QLQ-BN20; measured during screening, at response assessment II, and with beginning of RA III every 12 months until end of follow-up

OTHER OUTCOMES:
Comparison of de-escalated regimen to standard induction therapy regarding safety | up to 60 days after ASCT
  incidence of (Serious) adverse events, laboratory parameters:WBC <2.500/µl and platelets <80.000/μl , vital signs: blood pressure (mmHg), heart rate (bpm)
Comparison of de-escalated regimen to standard induction therapy regarding neurotoxicity | up to 24 months after end of treatment
  MoCA (Montreal Cognitive Assesment) performed at screening, EOT and every 12 months until end of follow-up
Comparison of de-escalated regimen to standard induction therapy regarding neurotoxicity | up to 24 months after end of treatment
  WAIS III (Wechsler Adult Intelligence scale) counting test performed at screening, EOT and every 12 months until end of follow-up
Comparison of de-escalated regimen to standard induction therapy regarding neurotoxicity | up to 24 months after end of treatment
  WAIS III (Wechsler Adult Intelligence scale) subtest similarities and verbal fluency test performed at screening, EOT and every 12 months until end of follow-up
Comparison of de-escalated regimen to standard induction therapy regarding neurotoxicity | up to 24 months after end of treatment
  Trail Making Test A and B, performed at screening, EOT and every 12 months until end of follow-up
Comparison of de-escalated regimen to standard induction therapy regarding neurotoxicity | up to 24 months after end of treatment
  Brief Test of Attention performed at screening, EOT and every 12 months until end of follow-up
Comparison of de-escalated regimen to standard induction therapy regarding neurotoxicity | up to 24 months after end of treatment
  Hopkins Verbal Learning Test performed at screening, EOT and every 12 months until end of follow-up
Comparison of de-escalated regimen to standard induction therapy regarding neurotoxicity | up to 24 months after end of treatment
  Grooved Pegboard Test, performed at screening, EOT and every 12 months until end of follow-up
Comparison of de-escalated regimen to standard induction therapy regarding neurotoxicity | up to 24 months after end of treatment
  Rey-Osterrieth-Complex-Figure-Test performed at screening, EOT and every 12 months until end of follow-up
Unplanned hospital admissions | up to 6 months after EOT visit
  Defined as in-patient hospitalization from randomization until 6 months after EOT visit (excluding those for study therapy and/or assessments, placement of an indwelling catheter, social/convenience admissions, respite care, elective or pre-planned treatment/surgery)
Length of hospital stays | up to 6 months after EOT visit
  Measured as number of nights in hospital from randomization and until 6 months after EOT. Hospitalization must be in relation to the disease or the administered treatment or due to toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Illerhaus, Prof, Principal Investigator — Klinikum Stuttgart
Locations (1):
- Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
After approval through ethics committee publication of study protocol. Anonymised patient data can be provided upon project related request.
Supporting Information: Study Protocol
Time Frame: Study protocol: 1st quarter 2021 Not before 2nd quarter 2028: Anonymised patient data
Access Criteria: To get access to anonymised patient data, a research proposal/project plan is required.